CLINICAL TRIAL: NCT04938271
Title: A Telemedicine Home-Based Study of Healables Wearable Electroceutical & Sports Sleeve Designed for Pain Relief & Improved Function in Mild to Moderate Knee Osteoarthritis Including in Persons With Chronic Illness Following Sports Injury
Brief Title: A Telehealth Study of a Wearable Electroceutical & Sports Sleeve for Knee Osteoarthritis Pain Relief & Improved Function
Acronym: HEAL01WMCOA1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Healables Ltd. (Industry)
Collaborators: Wolfson Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HEALABLES HEAL-01; IIA-71927 (Other Grant/Funding Number: Israel Innovation Authority); 0187-19-WOMC (Other: Edith Wolfson Medical Center, Holon, Israel)
Record Dates: First submitted 2021-05-30; First posted 2021-06-24 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Osteoarthritis, Knee
Keywords: osteoarthritis; wearable; electroceutical; telemedicine; microcurrent; medical device; pain relief; knee dysfunction; smart textile; e-textile; Telehealth; App; iPhone; smartphone; remote treatment; sports injury
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Alzheimer Disease; Athletic Injuries

STUDY DESIGN:
Intervention Model Description: Open label telemedicine home-based study to ascertain the potential effects of an App-driven wearable microcurrent electroceutical docked with an e-textile sports sleeve to relieve pain and improve function in subjects with mild to moderate knee arthritis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healables Wearable Microcurrent Electroceutical HEAL-122 with e-Textile Sports Sleeve (Experimental): Subjects activate electroceutical at home for 60 minutes (+/- 20 minutes) daily, 5 times per week, for 4 weeks
  Interventions: Device: HEAL-122 microcurrent electroceutical with e-textile sports knee sleeve

INTERVENTIONS:
Device: HEAL-122 microcurrent electroceutical with e-textile sports knee sleeve — Using a bluetooth connected iPhone, subject activates the HEAL-122 electroceutical device that is docked onto an e-textile sports knee sleeve worn on the osteoarthritic knee

SUMMARY:
The purpose of this telemedicine 24-person open-label study is to evaluate the safety and usability of a proprietary wearable microcurrent electroceutical (a device that delivers micro-ampere electronic pulses) made by Healables, Ltd. to promote healing of chronic mild to moderate knee osteoarthritis as shown by decreased disability and relief of pain. In this study, subjects treat themselves at home once/day for an hour using a smart phone to activate the device worn on an e-textile sports knee sleeve. Microcurrent signals are transmitted from a device thru built in conductive pathways to strategic electrodes placed above and below the knee. A proprietary App both activates therapeutic protocols to transmit microcurrent signals as well as allows user-generated recording of the status of knee pain & function prior to and following each treatment. These records are then transmitted to health professionals using software compliant with human use data transmission regulations including subject anonymity.

The rationale that the device would be effective is supported by microcurrent treatment for osteoarthritis at several US clinics including the prestigious Cleveland Clinic as well as by data of published randomized controlled clinical trials. One reason that more persons do not avail themselves of microcurrent therapy is that treatment usually requires several trips to a clinic often requiring considerable travel by a patient who may be in considerable pain. The health provider typically administers therapy in a clinic using electrodes with a desktop sized instrument. Our miniaturization of a microcurrent device and its use with wearable e-textiles such as a knee compression sleeve is a distinct advantage that enables regular use of effective therapy in home-based self-treatment to provide pain relief and improved knee function.

Microcurrent electrotherapy represents a significant improvement in pain control and healing since it employs current in the microampere range, 1000 times less than that of Transcutaneous Electrical Nerve Stimulator (TENS) devices that transmit millicurrent electrical signals. This study is designed to demonstrate use of a wearable microcurrent electroceutical at home for subjects to self-treat at their leisure in a comfortable environment that facilitates healing. Moreover, data communication via a smart phone App to health providers enables digital telemedicine for rapid collation and interpretation of relevant data.

DETAILED DESCRIPTION:
INTRODUCTION Definitions: an electroceutical, compared to a pharmaceutical, is a device that provides treatment by delivering potentially therapeutic electrical pulses; a microcurrent electroceutical delivers electrical pulses in the micro-ampere range and is distinguished from devices that deliver millicurrent which are electrical pulses in the milliampere range, 1000-fold greater than the micro ampere range.

Electrical microcurrent therapy represents a significant improvement in rapid pain control and acceleration of healing since it not only avoids the side effects of drugs including opioids and NSAIDs, but is also a superior electroceutical modality since it uses 1000-fold less electric current than that of Transcutaneous Electrical Nerve Stimulation (TENS), which requires application of current in the millicurrent range and can itself be painful and damaging to nerve tissues.

Electrotherapy, especially microcurrent electrical therapy, has been used to treat a variety of clinical conditions and is routinely used at pain clinics in the USA, most notable among them, the Cleveland Clinic, consistently rated among the top 3 medical centers in the USA. Microcurrent electro-therapy may be the best treatment for many pain-related disorders, since it not only provides fast relief of symptoms and promotes quick healing but also it has significantly fewer adverse side effects than many analgesic drugs. Indeed, this Cleveland Clinic website lists multiple diseases and disorders amenable to microcurrent therapy to ameliorate pain as do numerous published studies. Unfortunately, such microcurrent therapy is traditionally administered using a large desktop instrument through electrodes positioned by a health practitioner so that current can flow between the electrodes through the affected area of pain. While many practitioners in the USA are competent to administer such microcurrent therapy in both small and large clinical settings, treatment often requires significant travel by the patient who may be in considerable pain. Hence, patients frequently forego microcurrent therapy to avoid multiple trips to the health care provider at a clinic which may be quite distant.

Microcurrent Electroceutical: Healables Ltd. has determined that microcurrent therapy can be designed as a wearable medical device for use at home, at work or when travelling. This functional innovation provides a solution to provide widespread availability of microcurrent therapy. Healables has miniaturized a device that can deliver microcurrent electrotherapy and has devised a way to dock it to wearable e-textiles such sleeves, socks or body shirts with built in electrode paths to deliver microcurrent signals to the affected areas. Powered by an smart phone App (provided), the subject can wear the Healables device at home, work or in transit to provide timely and, if warranted, frequent microcurrent therapy at his/her leisure. Moreover, the App allows the subject to remotely communicate with health providers by digital health telecommunication to report and document daily progress.

The purpose of this clinical trial at the Edith Wolfson Medical Center (WMC) is to demonstrate the safety, tolerability and usability of a Healables electroceutical device in subjects with mild to moderate osteoarthritis pain and/or dysfunction to promote healing of chronic mild to moderate knee osteoarthritis as shown by relief of pain and decreased disability.

Microcurrent Putative Mechanisms of Action: Microcurrent electrical fields have been shown to stimulate cellular physiology and growth. In a preclinical study, microcurrent electric fields increased adenosine triphosphate (ATP) generation close to 500% whereas higher currents actually decreased the results. This study also demonstrated that microcurrent enhances amino acid transport and protein synthesis. In a clinical study, fibromyalgia pain was successfully treated with microcurrent therapy and pain improvement scores were accompanied by substantial reduction in serum inflammatory cytokines Interleukin-1 (IL-1), Interleukin-6 (IL-6), and tumor necrosis factor-alpha (TNF-α) levels as well as release of neuropeptide substance P and increases in serum Beta-endorphin and cortisol. This correlation indicated not only contributory treatment mechanisms effected by microcurrent therapy but also suggested that that such treatment can be objectively measured by observing changes in cytokines associated with pain and inflammation. Another suggested mechanism is based on the natural anti-oxidant ability of microcurrent to deliver electrons to tissues and saturate free radicals with required electrons. Such anti-oxidant activity is thought to repair local tissue damage that can be caused by a variety of chronic inflammatory illnesses including diabetes.

Study Design and Description This is a non-blinded, open label study. Subjects that have signed informed consent, have met all inclusion and none of the exclusion criteria will be enrolled in the study and treated. Each subject will be given an electroceutical device and a wearable knee sleeve that docks onto with the device and that shall be worn on the subject's leg with mild to moderate knee osteoarthritis. The subject is also provided with a smart phone phone (iPhone) with a proprietary App to run the device and data reporting software.

Subjects instructed by staff regarding device and App function and method of operation. Each treatment will comprise a self-treatment session at home of electroceutical microcurrent treatment for 60 +/- 20 minutes per day for 5 days per week for four consecutive weeks. Each treatment session will accompanied by use of the App to complete the 11-point Wong-Baker Visual Analog Scale (VAS) for knee pain prior to and following each treatment. The subject will also use the App once per week, every week of active treatment during the 1st 4 weeks of the study to score the 5-point, 12 question Knee Injury and Osteoarthritis Outcome Score (KOOS-12) for knee pain and dysfunction. In addition, for a 4-week follow up period after the 4 week treatment period, subjects will use the VAS and KOOS-12 weekly to assess residual effects of the treatments received during the 4 weeks of active treatment.

In addition to the periodic questionnaires completed by the subject using the App, the International Knee Documentation Committee (IKDC) questionnaire will be administered at the Wolfson Medical Center (WMC) osteoarthritis clinic at baseline and at weeks 2, 4 and 8. In this manner assessment will be made during active treatment, at the end of 4 weeks treatment and 4 weeks after the end of treatment to assess any residual effects of treatment after treatment has ended. The IKDC will be the primary goal to assess the effect of treatment on the level of pain and functionality of the subject's osteoarthritic knee.

Clinical Data Management Workflow Clinical data will be entered digitally from three sources. In the clinic the health practitioners will enter information into a tablet or other computer device that will transmit data to a Flaskdata backend. Such data will include the IKDC form and all info of the eCRF (electronic case report form). Another sources of data include data directly transmitted to Flaskdata from the device including, for example, measures of impedance, specific protocols used as well as times and lengths of use. A third component of data will be generated by subject responses to program queries and transmitted to Flaskdata via the App including questions regarding hydration and the Wong/Baker VAS pain levels and the 12-question KOOS-12 questionnaires described above.

All data from both the App as well as from the WMC clinic will be referred electronically to the health portals of Flaskdata.io to be securely and privately kept with de-identification according to the prerequisites of HIPPA and Good Clinical Practice (GCP). Data will be available to the WMC health professionals to monitor the subject's progress and use of the device and the App.

Treatment and reporting data from the App completed by the subject and from the e-CRFs (Electronic Case Report Forms) completed by WMC health providers also will be transmitted electronically to a database via Flaskdata.io for subsequent analysis in a de-identified and HIPPA compliant manner.

ELIGIBILITY:
Inclusion Criteria:

1. Mild to moderate osteoarthritis with pain and/or dysfunction in one or both knees as defined as Kellgren-Lawrence grade 1-3 as defined by radiograph or arthroscopy
2. Signed informed consent
3. Ages: 18 - 80 years of both genders

Exclusion Criteria:

1. Pacemaker or any electrically active implant
2. Health concerns disclosed at screening interview history and physical including initial laboratory values that in the opinion of a study health professional would preclude participation including a serious metabolic, infectious, neoplastic, neurologic or psychiatric disease.
3. Persons who have had knee orthopedic surgery with the exception of arthroscopic surgery since previous arthroscopic surgery is not an exclusion criterion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-11-22 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Number of device related serious adverse events recorded from baseline to end of study | baseline to end of study (8 weeks)
  The number of device related serious adverse events that occur in each subject during the entire eight weeks of the study including both the four weeks of active treatment as well as during the four weeks following treatment when potential residual effects of treatment will be observed.
Number of Subjects with Device Treatment-Related Effects on Knee Pain and Dysfunction as Measured by Changes from Baseline to 4 week End of Treatment in the International Knee Documentation Committee (IKDC) Osteoarthritis Index | Measured comparing changes from baseline to the end of 4 weeks
  Measurements of the International Knee Documentation Committee (IKDC) Osteoarthritis Index will be recorded by the investigator at the clinic at baseline and at the 4 week end of active treatment period. IKDC contains 10 questions; scoring 0 to 87 points in total (0 is worst and 87 is best). Study is intended to compare IKDC score between the 2 time points to determine possible improvement of worsening during the 4 week active treatment period.

SECONDARY OUTCOMES:
Number of Subjects with Device Treatment-Related Effects on Knee Pain and Dysfunction as Measured by Changes from Baseline through the 4 week End of Treatment Period using the 12-Question Knee Injury and Osteoarthritis Outcome Score (KOOS-12) | Measured comparing changes from baseline to the end of 4 weeks
  Measurements using the 12 question Knee injury and Osteoarthritis Outcome Score (KOOS-12) for knee pain and dysfunction will be recorded at baseline and weekly to the end of the 4 week active treatment period by each subject at home using a smart phone application (App) displaying a 5-point scale (0 to 4 points) for each of the 12 questions. In this scale, a higher number represents a worse outcome.
Number of Subjects with Device Treatment-Related Effects on Knee Pain as Measured by Changes from Baseline to the 4 week End of Treatment Period in the Wong-Baker Visual Analog Scale (VAS) | Measured comparing changes from baseline to the end of 4 weeks
  Measurements using the Wong-Baker Visual Analog Scale (VAS) for knee pain will be recorded at baseline and prior to and after each treatment during the 4 week active treatment period by each subject at home using a smart phone application (App) that displays the 11-point scale (0 to 10 points) VAS scale. In this scale, a higher number represents a worse outcome.

OTHER OUTCOMES:
Number of Subjects with Device Treatment-Related Effects on Knee Pain and Dysfunction as Measured by Changes from Baseline to 8 weeks End of the Study in the International Knee Documentation Committee (IKDC) Osteoarthritis Index | Baseline to 8 week visit end of study
  Measurements of the International Knee Documentation Committee (IKDC) Osteoarthritis Index will be recorded by the investigator at the clinic at baseline and at the 8 week end of the study. IKDC contains 10 questions; scoring 0 to 87 points in total (0 is worst and 87 is best). Study is intended to compare IKDC score between the 2 time points to determine possible improvement of worsening during the study comparing changes from the baseline to the 8 week end of the study.
Number of Subjects with Device Treatment-Related Effects on Knee Pain and Dysfunction as Measured by Changes from Baseline through the 8 week End of the Study using the 12-Question Knee Injury and Osteoarthritis Outcome Score (KOOS-12) | Measured comparing changes from baseline to the end of 8 weeks
  Measurements using the 12 question Knee injury and Osteoarthritis Outcome Score (KOOS-12) for knee pain and dysfunction will be recorded at baseline and weekly to the study end at 8 weeks by each subject at home using a smart phone application (App) displaying a 5-point scale (0 to 4 points) for each of the 12 questions. In this scale, a higher number represents a worse outcome. Study is intended to compare KOOS-12 score between the 2 time points to determine possible improvement of worsening during during the study comparing changes from the baseline to the 8 week end of the study.
Number of Subjects with Device Treatment-Related Effects on Knee Pain as Measured by Changes from Baseline through the 8 Weeks End of the Study in the Wong-Baker Visual Analog Scale (VAS) | Measured comparing changes from baseline to the end of 8 weeks
  Measurements using the Wong-Baker Visual Analog Scale (VAS) for knee pain will be recorded at baseline and, after the end of the 4 week active treatment period, weekly during the 4 week follow-up period to the end of week 8, by each subject at home using a smart phone application (App) that displays the 11-point scale (0 to 10 points) VAS scale. In this scale, a higher number represents a worse outcome. Study is intended to compare the VAS score between the 2 time points to determine possible improvement of worsening during during the study comparing changes from the baseline to the 8 week end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Hadar Oz, MD, Principal Investigator — Edith Wolfson Medical Center
Locations (1):
- Edith Wolfson Medical Center, Holon, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zizic TM, Hoffman KC, Holt PA, Hungerford DS, O'Dell JR, Jacobs MA, Lewis CG, Deal CL, Caldwell JR, Cholewczynski JG, et al. The treatment of osteoarthritis of the knee with pulsed electrical stimulation. J Rheumatol. 1995 Sep;22(9):1757-61. PMID 8523357
- [Background] Trock DH, Bollet AJ, Dyer RH Jr, Fielding LP, Miner WK, Markoll R. A double-blind trial of the clinical effects of pulsed electromagnetic fields in osteoarthritis. J Rheumatol. 1993 Mar;20(3):456-60. PMID 8478852
- [Background] Curtis D, Fallows S, Morris M, McMakin C. The efficacy of frequency specific microcurrent therapy on delayed onset muscle soreness. J Bodyw Mov Ther. 2010 Jul;14(3):272-9. doi: 10.1016/j.jbmt.2010.01.009. Epub 2010 Feb 19. PMID 20538225
- See also: Use of microcurrent treatment for many disorders including arthritis at the Cleveland Clinic — http://my.clevelandclinic.org/health/treatments/15935-frequency-specific-microcurrent